CLINICAL TRIAL: NCT00863265
Title: Regulation of Cholesterol Absorption: LDL Cholesterol Response to a Combination of Phytosterols and Ezetimibe (Phyto-3)
Brief Title: Phytosterols, Ezetimibe, and Cholesterol Metabolism
Acronym: Phyteaux-III
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Utah State University (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: CANUSU-phyto3; R01HL050420 (NIH)
Record Dates: First submitted 2009-03-16; First posted 2009-03-17 (Estimated); Results first posted 2018-06-01 (Actual); Last update posted 2018-06-01 (Actual); Status verified 2018-05

CONDITIONS: Hypercholesterolemia; Coronary Heart Disease
Keywords: Phytosterols; Ezetimibe; Cholesterol Excretion; Cholesterol Absorption; Diet; Mass Spectrometry; Deuterium
MeSH Terms: conditions — Hypercholesterolemia; Coronary Disease | interventions — Ezetimibe; Phytosterols

STUDY DESIGN:
Intervention Model Description: This is a randomized, crossover design. There are three periods of 21 days separated by two 7 day washouts. All subjects eat a controlled low-phytosterol diet for each of the three periods. During period B placebo phytosterols and placebo ezetimibe are given. During period C phytosterol placebo and active ezetimibe are given. During period A active phytosterols and active ezetimibe are given. Periods are assigned in random order as described in Arms below.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Phytosterols solutions were provided as food oil only (placebo) or food oil containing 2000 mg/day phytosterols (Phytosterols). Active and placebo ezetimibe tablets were provided by Merck.
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Crossover order ABC (Experimental): The order of treatments is A (phytosterols + ezetimibe), B (double placebo), and C (active ezetimibe and phytosterol placebo).
  Interventions: Drug: Ezetimibe; Other: Phytosterols + ezetimibe; Other: Placebo
- Crossover order BCA (Experimental): The order of treatments is B (double placebo), C (active ezetimibe and phytosterol placebo), and A (phytosterols + ezetimibe).
  Interventions: Drug: Ezetimibe; Other: Phytosterols + ezetimibe; Other: Placebo
- Crossover order BAC (Experimental): The order of treatments is B (double placebo), A (phytosterols + ezetimibe), and C (active ezetimibe and phytosterol placebo)
  Interventions: Drug: Ezetimibe; Other: Phytosterols + ezetimibe; Other: Placebo
- Crossover order ACB (Experimental): The order of treatments is A (phytosterols + ezetimibe), C (active ezetimibe and placebo phytosterols, and B (double placebo).
  Interventions: Drug: Ezetimibe; Other: Phytosterols + ezetimibe; Other: Placebo
- Crossover order CAB (Experimental): The order of treatments is C (active ezetimibe and placebo phytosterols), A (phytosterols + ezetimibe), and B (double placebo).
  Interventions: Drug: Ezetimibe; Other: Phytosterols + ezetimibe; Other: Placebo
- Crossover order CBA (Experimental): The order of treatments is C (active ezetimibe and placebo phytosterols), B (double placebo), and A (phytosterols and ezetimibe).
  Interventions: Drug: Ezetimibe; Other: Phytosterols + ezetimibe; Other: Placebo

INTERVENTIONS:
Drug: Ezetimibe — Subjects will undergo three diet periods of 21 days each separated by 7 day washouts. Food will be supplied by a metabolic kitchen and will consist of a phytosterol-deficient baseline diet. During each period subjects will receive either phytosterol esters or placebo and ezetimibe or placebo.
  Other Names: C
Other: Phytosterols + ezetimibe — Subjects will undergo three diet periods of 21 days each separated by 7 day washouts. Food will be supplied by a metabolic kitchen and will consist of a phytosterol-deficient baseline diet. During each period subjects will receive either phytosterol esters or placebo and ezetimibe or placebo.
  Other Names: A
Other: Placebo
  Other Names: B

SUMMARY:
Phytosterols and ezetimibe each reduce intestinal cholesterol absorption by 30-55% but appear to have different mechanisms of action. The investigators' hypothesis is that phytosterols and ezetimibe given together will block cholesterol absorption in an additive fashion. In a randomized, placebo-controlled crossover trial the effects of placebo, ezetimibe treatment and ezetimibe plus phytosterol treatment will be measured.

DETAILED DESCRIPTION:
The investigators will perform a randomized, placebo-controlled crossover feeding study in 25 subjects with greater than ideal levels of LDL cholesterol who do not require anti-cholesterol drug treatment. Subjects will consume a baseline diet provided by a feeding center that is deficient in phytosterols for three periods of 21 days separated by 7-day washout periods. Treatments will be given in random order During period B placebo phytosterols and placebo ezetimibe will be given; during period C placebo phytosterols and active ezetimibe will be given; during period A active phytosterols and active ezetimibe will be given. Study endpoints are fecal cholesterol excretion and percent cholesterol absorption determined by gas chromatography/mass spectrometry and circulating LDL cholesterol.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of any race or ethnicity between 18 to 80 years of age;
* Body mass index between 20 - 35 kg/m2;
* LDL-cholesterol between 130 - 189 mg/dL based on the average of duplicate screening measures. If the two LDL-C levels differ by more than 30 mg/dL, a third test will be scheduled with all three results averaged;
* Free of chronic disease;
* Willing to eat only the foods that are provided by the Center during the diet periods;
* Willing to abstain from the consumption of alcohol for 48-hours prior to blood draw days;
* Willing to drink no more than 5 cups of caffeine-containing beverages a day.

Exclusion Criteria:

* Age < 18 or > 80 years;
* Based on duplicate screening laboratory values: 1)LDL-C >=190 mg/dL; 2)TG >=250 mg/dL;3)blood pressure >= 160 mm Hg systolic or 95 mm Hg diastolic;
* Documented presence of atherosclerotic disease;
* Diabetes mellitus;
* Renal, hepatic, endocrine, gastrointestinal, hematological or other systemic disease;
* Body mass index > 35;
* For women, pregnancy, breast feeding or postpartum < 6 months;
* For women, peri-menopausal;
* For women, sexually active but not practicing effective birth control methods;
* History of drug or alcohol abuse;
* History of depression or mental illness requiring treatment or medication within the last 6 months;
* multiple food allergies or significant food preferences or restrictions that would interfere with diet adherence;
* Chronic use of over-the-counter medication which would interfere with study endpoints including laxatives and antacids;
* Lifestyle or schedule incompatible with the study protocol;
* Planned continued use of dietary supplements through the study trial;
* Taking any lipid-lowering, or other medications known to affect blood cholesterol.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2009-06; Primary Completion 2009-10 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Ostlund, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Center for Advance Nutrition at Utah State University, Logan, Utah, United States

REFERENCES:
- [Result] Lin X, Racette SB, Lefevre M, Ma L, Spearie CA, Steger-May K, Ostlund RE Jr. Combined effects of ezetimibe and phytosterols on cholesterol metabolism: a randomized, controlled feeding study in humans. Circulation. 2011 Aug 2;124(5):596-601. doi: 10.1161/CIRCULATIONAHA.110.006692. Epub 2011 Jul 18. PMID 21768544

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 175 subjects were screened and 153 were excluded prior to randomization. 75 did not meet screening criteria, 39 declined to participate and 39 were not able to perform functions needed for the study. 22 Subjects were randomized and 21 completed the study.
Groups:
- Crossover Order ABC; Crossover Order BCA; Crossover Order BAC; Crossover Order ACB; Crossover Order CAB; Crossover Order CBA: Subjects will undergo 3 periods of 21 days on a controlled diet plus phytosterols/placebo and ezetimibe/placebo. A washout of 7 days occurs between periods.
  A. Phytosterols 2000 mg/day and ezetimibe 10 mg/day. B. Phytosterol placebo and ezetimibe placebo. C. Phytosterol placebo and active ezetimibe 10 mg/day. ezetimibe plus phytosterols.
Period: Overall Study
Arm/Group | Crossover Order ABC | Crossover Order BCA | Crossover Order BAC | Crossover Order ACB | Crossover Order CAB | Crossover Order CBA
Started | 4 | 3 | 4 | 4 | 4 | 3
Completed | 4 | 3 | 4 | 4 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: All study participants.
Arm/Group | All Study Participants
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  race: white | 20
  race: asian | 1
  race: hispanic | 1

OUTCOME MEASURES:

1. Primary Outcome: Cholesterol Excretion
Description: Milligrams of fecal cholesterol and cholesterol metabolites excreted per day
Time Frame: At the end of week 3 on each diet
Population: Healthy subjects
Measure: Mean (95% Confidence Interval); unit: mg per day
Groups:
- Phytosterol-Deficient Diet: Phytosterol-deficient diet plus ezetimibe placebo plus phytosterol placebo.
  Phytosterol-Deficient Diet, Ezetimibe 10 mg, Phytosterol Esters Containing 2000 mg Phytosterols: Subjects will undergo three diet periods of 21 days each. Food will be supplied by a metabolic kitchen and will consist of a phytosterol-deficient baseline diet. Subjects will also receive either no active treatment, ezetimibe, or ezetimibe plus phytosterols.
- Diet Plus Ezetimibe: Phytosterol-deficient diet plus 10 mg/day of ezetimibe plus phytosterol placebo.
  Phytosterol-Deficient Diet, Ezetimibe 10 mg, Phytosterol Esters Containing 2000 mg Phytosterols: Subjects will undergo three diet periods of 21 days each. Food will be supplied by a metabolic kitchen and will consist of a phytosterol-deficient baseline diet. Subjects will also receive either no active treatment, ezetimibe, or ezetimibe plus phytosterols.
- Diet Plus Ezetimibe Plus Phytosterols: Phytosterol-deficient diet plus 10 mg/day of ezetimibe plus 2000 mg/day of phytosterols.
  Phytosterol-Deficient Diet, Ezetimibe 10 mg, Phytosterol Esters Containing 2000 mg Phytosterols: Subjects will undergo three diet periods of 21 days each. Food will be supplied by a metabolic kitchen and will consist of a phytosterol-deficient baseline diet. Subjects will also receive either no active treatment, ezetimibe, or ezetimibe plus phytosterols.
Arm/Group | Phytosterol-Deficient Diet | Diet Plus Ezetimibe | Diet Plus Ezetimibe Plus Phytosterols
Number analyzed (Participants) | 21 | 21 | 21
mg per day | 505 [386 to 625] | 794 [615 to 973] | 962 [757 to 1168]
Statistical Analysis 1: Comparison: Phytosterol-Deficient Diet vs Diet Plus Ezetimibe; Phytosterol Diet compared to Ezetimibe; Test type: Equivalence; p = 0.01, ANOVA; Mean Difference (Final Values) = 289 — The estimation parameter is the difference between the placebo group and the ezetimibe group
Statistical Analysis 2: Comparison: Phytosterol-Deficient Diet vs Diet Plus Ezetimibe Plus Phytosterols; Placebo vs. Ezetimibe Plus Phytosterols; Test type: Equivalence — The hypothesis is that groups are equal; p < 0.01, ANOVA; Mean Difference (Final Values) = 457
Statistical Analysis 3: Comparison: Diet Plus Ezetimibe vs Diet Plus Ezetimibe Plus Phytosterols; Ezetimibe vs. Ezetimibe Plus Phytosterols; Test type: Equivalence — The hypothesis is that groups are equal; p < 0.01, ANOVA; Mean Difference (Final Values) = 168

2. Primary Outcome: Percent Cholesterol Absorption
Description: Percent of intestinal cholesterol absorbed. Intestinal cholesterol is comprised of dietary cholesterol intake and endogenous cholesterol secreted into the intestinal lumen. Cholesterol absorption is the percent of intestinal cholesterol that is taken back up into the body and excluded from fecal excretion. It is also referred to as the efficiency of intestinal cholesterol absorption.
Time Frame: Determined on the final 5 days of each dietary period
Measure: Mean (95% Confidence Interval); unit: Percent
Groups:
- Phytosterol-Deficient Diet: Phytosterol-deficient diet plus ezetimibe placebo plus phytosterol placebo
- Diet Plus Ezetimibe: Phytosterol-deficient diet plus ezetimibe plus phytosterol placebo
- Diet Plus Ezetimibe Plus Phytosterols: Phytosterol-deficient diet plus ezetimibe plus phytosterols
Arm/Group | Phytosterol-Deficient Diet | Diet Plus Ezetimibe | Diet Plus Ezetimibe Plus Phytosterols
Number analyzed (Participants) | 21 | 21 | 21
Percent | 69.0 [61.8 to 76.2] | 46.2 [38.5 to 53.9] | 32.6 [26.9 to 38.3]
Statistical Analysis 1: Comparison: Phytosterol-Deficient Diet vs Diet Plus Ezetimibe; The hypothesis is that groups are equal; Test type: Equivalence — Not applicable in this study; p < 0.01, ANOVA — Adjusted for multiple comparisons; Mean Difference (Final Values) = 22.8
Statistical Analysis 2: Comparison: Phytosterol-Deficient Diet vs Diet Plus Ezetimibe Plus Phytosterols; Placebo vs. Ezetimibe Plus Phytosterols; Test type: Equivalence; p < 0.01, ANOVA — Adjusted for multiple comparisons; Mean Difference (Final Values) = 36.4
Statistical Analysis 3: Comparison: Diet Plus Ezetimibe vs Diet Plus Ezetimibe Plus Phytosterols; The hypothesis is that groups are equal; Test type: Equivalence; p < 0.01, ANOVA — Adjusted for multiple comparisons; Mean Difference (Final Values) = 13.6

3. Primary Outcome: LDL Cholesterol
Time Frame: At the end of week 3 on each diet
Population: Healthy subjects
Measure: Mean (95% Confidence Interval); unit: mg/deciliter
Groups:
- Phytosterol-Deficient Diet Plus Ezetimibe: Phytosterol-Deficient Diet Plus Ezetimibe Plus Phytosterol Placebo.
- Phytosterol-Deficient Diet Plus Ezetimibe Plus Phytosterols: Phytosterol-deficient diet plus ezetimibe plus phytosterols.
Arm/Group | Phytosterol-Deficient Diet | Phytosterol-Deficient Diet Plus Ezetimibe | Phytosterol-Deficient Diet Plus Ezetimibe Plus Phytosterols
Number analyzed (Participants) | 21 | 21 | 21
mg/deciliter | 129 [116 to 142] | 108 [97 to 119] | 101 [90 to 112]
Statistical Analysis 1: Comparison: Phytosterol-Deficient Diet vs Phytosterol-Deficient Diet Plus Ezetimibe; The hypothesis is that groups are equal; Test type: Equivalence; p < 0.01, ANOVA; Mean Difference (Final Values) = 21
Statistical Analysis 2: Comparison: Phytosterol-Deficient Diet vs Phytosterol-Deficient Diet Plus Ezetimibe Plus Phytosterols; The hypothesis is that all groups are equal; Test type: Equivalence; p < 0.01, ANOVA — Adjusted for multiple comparisons; Mean Difference (Final Values) = 28
Statistical Analysis 3: Comparison: Phytosterol-Deficient Diet Plus Ezetimibe vs Phytosterol-Deficient Diet Plus Ezetimibe Plus Phytosterols; The hypothesis is that groups are equal; Test type: Equivalence; p < 0.05, ANOVA — Adjusted for multiple comparisons; Mean Difference (Final Values) = 7

ADVERSE EVENTS:
Arm/Group | Phytosterol-Deficient Diet | Diet Plus Ezetimibe | Diet Plus Ezetimibe Plus Phytosterols
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No